CLINICAL TRIAL: NCT06068179
Title: The Efficacy and Safety of Combining Mycophenolate Mofetil With Methimazole on Remission of Newly Diagnosis Graves' Disease (3M-RGD Trial): an Open-label, Randomized Trial
Brief Title: Graves' Disease Remission Study: MycoMeth Combo
Acronym: 3M-RGD
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: The First Affiliated Hospital of Xiamen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: XMFHIIT-2023SL059
Record Dates: First submitted 2023-09-28; First posted 2023-10-05 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2023-09

CONDITIONS: Graves' Disease
Keywords: Newly Diagnosed Graves' Disease; Mycophenolate Mofetil; Methimazole; Remission
MeSH Terms: conditions — Graves Disease | interventions — Mycophenolic Acid; Methimazole

STUDY DESIGN:
Intervention Model Description: Eligible patients will be randomly assigned to intervention group (Mycophenolate Mofetil combine with methimazole) or control group (methimazole standard therapy) for 12 months.
Who Masked: Outcomes Assessor
Masking Description: The study grouping will be blinded to outcomes assessor.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): Mycophenolate Mofetil 0.5 twice daily for 12 months added to methimazole standard therapy.
  Interventions: Drug: Mycophenolate Mofetil, Oral, 250 Mg; Drug: methimazole, oral, 10mg
- control group (Active Comparator): Methimazole 15-30mg daily initially, then titrate to maintenance dose. Beta-blocker used when necessary.
  Interventions: Drug: methimazole, oral, 10mg

INTERVENTIONS:
Drug: Mycophenolate Mofetil, Oral, 250 Mg — Mycophenolate Mofetil, Oral, 500Mg twice daily for 12 months, combined with methimazole standard therapy
  Arms: intervention group
Drug: methimazole, oral, 10mg — Methimazole 15-30mg daily initially then titrate to maintenance dose.

SUMMARY:
A randomized study to evaluate the efficacy and safety of combining mycophenolate mofetil with methimazole in patients with newly diagnosed Graves' disease.

DETAILED DESCRIPTION:
The remission rate of methimazole standard therapy in patients with newly diagnosed Graves' disease is only around 50%. Main reason for the low remission rate is methimazole therapy is not a drug targeting etiology of Graves' disease. The investigators hypothesize that adding mycophenolate mofetil, an immunosuppressor, to methimazole standard therapy will improve remission rate. The study will evaluate the efficacy and safety of combining mycophenolate mofetil with methimazole in patients with newly diagnosed Graves' disease. 205 eligible patients will be randomized to mycophenolate mofetil combined with methimazole therapy or methimazole standard therapy. The primary outcome is the remission rate at 12 months.

ELIGIBILITY:
Inclusion Criteria:

- 1. aged 18 to 60 years.

2. Patients newly diagnosed with Graves' disease.

Exclusion Criteria:

* 1. Patients with Graves' disease who have undergone treatment or experienced relapse.

  2. Hyperthyroidism due to other etiologies (toxic multinodular goiter, toxic thyroid adenoma, Hashimoto's thyroiditis, subacute thyroiditis, iodine-induced hyperthyroidism, etc.).

  3. Individuals requiring intervention for moderate to severe thyroid eye disease at the time of enrollment.

  4. Patients with hyperthyroidism requiring surgery due to concurrent thyroid cancer.

  5. Those with severe liver or kidney dysfunction (ALT or AST > 3 times the upper limit of normal reference values, blood creatinine > 135 mol/L for males, and 110 mol/L for females).

  6. Individuals with leukopenia (WBC < 3.0×109/L).

  7. Patients with severe heart failure (NYHA class III or IV).

  8. Individuals with chronic or severe infections such as pulmonary tuberculosis, hepatitis B, etc.

  9. Pregnant women, breastfeeding women, those planning pregnancy in the near future, or individuals who cannot comply with contraception during trial.

  10. Participants in or previously involved in other clinical studies.

  11. Individuals unwilling or unable to comply with follow-up or unwilling to participate.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 205 (Estimated)
Dates: Start 2023-10-16 (Actual); Primary Completion 2025-10-08 (Estimated); Study Completion 2026-10-08 (Estimated)

PRIMARY OUTCOMES:
Remission rate | 12 months
  Remission is defined as normal thyroid function, TRAb level at methimazole maintenance dose

CONTACTS AND LOCATIONS:
Overall Officials: Fangsen Xiao, MD, Principal Investigator — The first affiliated hospital of Xiamen University Medical College
Locations (1):
- Xiao Fangsen, Xiamen, Fujian, China

IPD SHARING:
Plan to Share IPD: No
No plan to share IPD

REFERENCES:
- [Result] Davies TF, Andersen S, Latif R, Nagayama Y, Barbesino G, Brito M, Eckstein AK, Stagnaro-Green A, Kahaly GJ. Graves' disease. Nat Rev Dis Primers. 2020 Jul 2;6(1):52. doi: 10.1038/s41572-020-0184-y. PMID 32616746
- [Result] Burch HB, Cooper DS. Management of Graves Disease: A Review. JAMA. 2015 Dec 15;314(23):2544-54. doi: 10.1001/jama.2015.16535. PMID 26670972
- [Result] Smith TJ, Hegedus L. Graves' Disease. N Engl J Med. 2016 Oct 20;375(16):1552-1565. doi: 10.1056/NEJMra1510030. No abstract available. PMID 27797318
- [Result] Kahaly GJ. Management of Graves Thyroidal and Extrathyroidal Disease: An Update. J Clin Endocrinol Metab. 2020 Dec 1;105(12):3704-20. doi: 10.1210/clinem/dgaa646. PMID 32929476
- [Result] Wiersinga WM. Graves' Disease: Can It Be Cured? Endocrinol Metab (Seoul). 2019 Mar;34(1):29-38. doi: 10.3803/EnM.2019.34.1.29. PMID 30912336
- [Result] Ross DS, Burch HB, Cooper DS, Greenlee MC, Laurberg P, Maia AL, Rivkees SA, Samuels M, Sosa JA, Stan MN, Walter MA. 2016 American Thyroid Association Guidelines for Diagnosis and Management of Hyperthyroidism and Other Causes of Thyrotoxicosis. Thyroid. 2016 Oct;26(10):1343-1421. doi: 10.1089/thy.2016.0229. PMID 27521067
- [Result] Torlinska B, Hazlehurst JM, Nirantharakumar K, Thomas GN, Priestley JR, Finnikin SJ, Saunders P, Abrams KR, Boelaert K. wEight chanGes, caRdio-mEtabolic risks and morTality in patients with hyperthyroidism (EGRET): a protocol for a CPRD-HES linked cohort study. BMJ Open. 2021 Oct 1;11(10):e055219. doi: 10.1136/bmjopen-2021-055219. PMID 34598995
- [Result] Broen JCA, van Laar JM. Mycophenolate mofetil, azathioprine and tacrolimus: mechanisms in rheumatology. Nat Rev Rheumatol. 2020 Mar;16(3):167-178. doi: 10.1038/s41584-020-0374-8. Epub 2020 Feb 13. PMID 32055040
- [Result] Prussick L, Plotnikova N, Gottlieb A. Mycophenolate Mofetil in Severe Atopic Dermatitis: A Review. J Drugs Dermatol. 2016 Jun 1;15(6):715-8. PMID 27272078
- [Result] Barbesino G, Salvi M, Freitag SK. Future Projections in Thyroid Eye Disease. J Clin Endocrinol Metab. 2022 Aug 8;107(Suppl_1):S47-S56. doi: 10.1210/clinem/dgac252. PMID 36346684
- [Result] Kahaly GJ, Riedl M, Konig J, Pitz S, Ponto K, Diana T, Kampmann E, Kolbe E, Eckstein A, Moeller LC, Fuhrer D, Salvi M, Curro N, Campi I, Covelli D, Leo M, Marino M, Menconi F, Marcocci C, Bartalena L, Perros P, Wiersinga WM; European Group on Graves' Orbitopathy (EUGOGO). Mycophenolate plus methylprednisolone versus methylprednisolone alone in active, moderate-to-severe Graves' orbitopathy (MINGO): a randomised, observer-masked, multicentre trial. Lancet Diabetes Endocrinol. 2018 Apr;6(4):287-298. doi: 10.1016/S2213-8587(18)30020-2. Epub 2018 Jan 31. PMID 29396246
- [Result] Rajabi MT, Rafizadeh SM, Mohammadi A, Eshraghi B, Mohammadi N, Hosseini SS, Rajabi MB, Keshmirshekan MM, Shahriari M, Poursayed Lazarjani SZ, Parandin MM. Mycophenolate Mofetil (CellCept(R)) in Combination With Low Dose Prednisolone in Moderate to Severe Graves' Orbitopathy. Front Med (Lausanne). 2022 Feb 11;9:788228. doi: 10.3389/fmed.2022.788228. eCollection 2022. PMID 35223896
- [Result] Feng W, Hu Y, Zhang C, Shi H, Zhang P, Yang Y, Chen S, Cui W, Cui D. Efficacy and safety of mycophenolate mofetil in the treatment of moderate to severe Graves' orbitopathy: a meta-analysis. Bioengineered. 2022 Jun;13(6):14719-14729. doi: 10.1080/21655979.2022.2101191. PMID 35959915